CLINICAL TRIAL: NCT07067788
Title: A Clinical Comparison of Siemens Mammomat B.Brilliant , A Novel Wide-Angel Digitial Breast Tomosynthesis System With Siemens Mammomat Revelation , A Standard Wide-Angle Digital Breast Tomosynthesis System
Brief Title: B.Brilliant Revelation Comparision Study
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Siemens Corporation, Corporate Technology (Industry)
Responsible Party: Sponsor
Other Study IDs: 857586
Record Dates: First submitted 2025-05-12; First posted 2025-07-16 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer Screening
Keywords: breast; mammogram; breast cancer; female
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Breast imaging in Females: Females who are equal to or greater than 18 years of age are scheduled to have additional imaging due to findings of calcifications or lesions with calcifications on a screening mammogram.
  Interventions: Diagnostic Test: Breast Imaging

INTERVENTIONS:
Diagnostic Test: Breast Imaging — Intervention using an FDA-approved mammogram machine.

SUMMARY:
This is an observational study to evaluate the MAMMOMAT B.brilliant system. All diagnostic decisions are made by the treating radiologist based upon standard of care clinical imaging acquired on FDA approved devices

DETAILED DESCRIPTION:
Women scheduled at Pennsylvania Hospital to undergo a standard of care diagnostic imaging exam after having had a standard of care screening exam performed on either the MAMMOMAT B.brilliant (NDBT) or the MAMMOMAT Revelation (DBT) mammography system with findings consistent with suspicious calcifications or calcifications associated with other lesion types will be eligible and approached to enroll in the study. Participants must be ≥ 18 years of age. Up to 125 evaluable participants will be enrolled.

Eligible and consented participants enrolled in the study will receive standard of care diagnostic imaging on the same mammography system as the screening exam and receive two additional research images on the other mammography system.

Both mammographic units are FDA approved and located at Pennsylvania Hospital.

The research scans required for this study will include either 5-8 seconds or 25 seconds of compression in two views (MLO & CC) of the affected breast (breast with suspicious calcifications at screening). Data will be collected to evaluate image quality regarding the visibility of calcifications. This study seeks to evaluate MAMMOMAT B.brilliant, which has decreased acquisition time and increased conspicuity of calcifications, as a replacement to standard wide-angle imaging as on the MAMMOMAT Revelation.

This is an observational study to evaluate the MAMMOMAT B.brilliant system. All diagnostic decisions are made by the treating radiologist based upon standard of care clinical imaging acquired on FDA approved devices

ELIGIBILITY:
Inclusion Criteria

1. Participants will be ≥ 18 years of age.
2. Participants will be females (sex assigned at birth).
3. Participants will be presenting for clinical diagnostic mammography with suspicious calcifications or calcifications associated with other lesion types
4. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria

1. Females who are breast-feeding will not be eligible for this study
2. Pregnant women will not be included. All females of childbearing potential must attest that they are not pregnant.
3. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician.
4. Any current medical condition, illness, or disorder, as assessed by medical record review and/or self-reported, that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — females whose gender is assigned at birth.
Study Population: Women are coming back for diagnostic imaging, whose screening mammogram shows findings of calcifications or lesions with calcifications, who are equal to or greater than 18 years of age.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of two Siemen System B.brillant and the Revelation | From enrollment to the end of study at 18 months
  • To assess whether the MAMMOMAT B.brilliant, a Novel Wide-Angle Digital Breast Tomosynthesis (NDBT) System, leads to better visualization of calcifications compared to the MAMMOMAT Revelation, a standard wide-angle Digital Breast Tomosynthesis (DBT) System, including the assessment of calcifications on synthetic images for both tomosynthesis scans.

SECONDARY OUTCOMES:
Accuracy of Calcifications and patient survey | From enrollment to the end of study at 18 months
  • To evaluate the accuracy of B.brilliant for predicting the number of calcifications and extent of the calcification cluster(s) and morphology compared to standard wide-angle DBT (including synthetic images for both) with diagnostic magnification views as the gold standard.
Assessing the pain on two standard mammogram scanners | From enrollment to the end of study at 18 months
  To assess whether subjects imaged with B.brilliant and standard wide-angle DBT perceive any difference in ease of exam or pain. We are using a numerical pain scale, a 0 to 5 point scale. 0 no pain and 5 severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Brian S Englander, MD, Principal Investigator — Pennsylvania Hospital
Locations (1):
- Pennsylvania Hospital, Center for Breast Imaging, Philadelphia, Pennsylvania, United States